CLINICAL TRIAL: NCT01990755
Title: Lack of Efficacy of Psychological and Pharmacological Treatments of Eating Disorders: Neurobiological Background
Brief Title: Neurobiology of Eating Disorders Treatments
Acronym: NEDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Federico Amianto, Dottor, University of Turin, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brambilla trial
Record Dates: First submitted 2013-09-24; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa | interventions — Cognitive Behavioral Therapy; Olanzapine; chlordesmethyldiazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT (Cognitive Behavioral Therapy) (Active Comparator): Investigates the effects of cognitive-behavioral therapy (CBT), on the secretion of brain dopamine (DA), noradrenalin (NE) and serotonin (5-HT) in a group of 50 female inpatients, 14 with AN restricter type (AN-R), 14 with the bingeing-purging type (AN-BP), and 22 with BN.
  Associated intervention (non of interest): psychiatric management (with tranquillizer: delorazepam), nutritional rehabilitation
  Interventions: Behavioral: CBT (Cognitive Behavioral Therapy); Dietary Supplement: nutritional rehabilitation; Drug: delorazepam
- IBPP (IP brief psychotherapy ) (Active Comparator): Investigates the effects in 15 AN and 17 BN patients of an individual psychology brief psychotherapy (IBPP) on psychological alterations and DA secretion measured as peripheral blood values of HVA before and after treatment.
  Associated intervention (non of interest): psychiatric management (with tranquillizer: delorazepam), nutritional rehabilitation.
  Interventions: Other: IBPP (individual psychology brief psychotherapy); Dietary Supplement: nutritional rehabilitation; Drug: delorazepam
- CBT + OLANZAPINE (5 MG) (Active Comparator): The study evaluated in 18 AN-R and 12 AN-BP patients the effects of CBT and of CBT associated with orally administered 5 mg olanzapine on the psychopathological aspects of the disease and on the secretion of HVA.
  Associated intervention (non of interest): psychiatric management (with tranquillizer: delorazepam), nutritional rehabilitation
  Interventions: Drug: CBT + OLANZAPINE; Dietary Supplement: nutritional rehabilitation; Drug: delorazepam

INTERVENTIONS:
Behavioral: CBT (Cognitive Behavioral Therapy) — It is a worldwide known form of psychotherapy for eating disorders
  Arms: CBT (Cognitive Behavioral Therapy)
Other: IBPP (individual psychology brief psychotherapy) — It is a worldwide known form of psychotherapy for eating disorders
  Other Names: B-APP: brief adlerian psychodynamic psychotherapy
  Arms: IBPP (IP brief psychotherapy )
Drug: CBT + OLANZAPINE — It is a worldwide known form of psychotherapy for eating disorders associated with a new antipsychotic with good efficacy on anorexia nervosa
  Arms: CBT + OLANZAPINE (5 MG)
Dietary Supplement: nutritional rehabilitation — all patients were followed-up monthly with nutritionist and dietitian visits
Drug: delorazepam — all patients were followed-up with psychiatric visits with symptomatic drug administration (tranquillizer: delorazepam) where necessary

SUMMARY:
Background. Treatments of eating disorders result too often in partial psychological and physical remission, chronic course, dropout, relapse and death, with no fully known explanations for this failure. In order to clarify this problem, we conducted a three branches study to identify the biochemical background of cognitive-behavioral psychotherapy (CBT), individual psychology brief psychotherapy (IBPP), and psychotherapy-pharmacotherapy with CBT+olanzapine in anorexics (AN) and bulimics (BN) by measuring the levels of plasma homovanillic acid (HVA) for dopamine secretion, plasma 3-methoxy-4-hydroxy-phenylglycol (MHPG) for noradrenalin secretion, and platelet [3 Hydrogen]-Paroxetine-binding Bmax and Kd for serotonin transporter function. The data were then compared with psychopathological and physical alterations. Methods. Branch 1 investigated the effects of 4 months of CBT on plasma HVA, MHPG and [3 Hydrogen]-Par-binding in 14 AN-restricted, 14 AN-bingeing/purging, and 22 BN inpatients. Branch 2 investigated the effects of 4 months of IBPP on plasma HVA in 15 AN and 17 BN outpatients. Branch 3 investigated the effect of 3 months of CBT+olanzapine (5 mg/day) in 30 AN outpatients. The data are analyzed using one-way ANOVA for repeated measures for the changes between basal and post-treatment biological and psychological parameters, two-way ANOVA for repeated measures for the differences in the psychobiological data in the 3 groups, Spearman's test for the correlations between basal and final changes in the psychological and biological scores.

ELIGIBILITY:
Inclusion Criteria:

* eating disorders full diagnosis according to Diagnostic and Statistical Manual (DSM-IV)
* age between 15 and 35
* female gender

Exclusion Criteria:

* associated major psychiatric problems
* mental retardation

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change in brain secretion of Dopamine at 6 months | 6 months
  plasma homovanillic acid (HVA) measured before and after the therapeutic intervention in each branch.
change in brain secretion of Noradrenaline at 6 months | 6 months
  plasma 3-methoxy-4-hydroxyphenylglycol (MHPG) measured before and after the therapeutic intervention in each branch
change in brain secretion of serotonin at 6 months | 6 months
  the platelet paroxetine binding ([3 Hydrogen]-Par-binding): Bmax (maximum binding capacity) and Kd (dissociation constant) measured before and after the therapeutic intervention in each branch.

SECONDARY OUTCOMES:
Eating Psychopathology improvement after treatments at 6 months | 6 months
  Eating Disorders Examination-12 (EDE 12)
Depressive Psychopathology improvement after 6 months | 6 months
  Beck Depression Inventory (BDI)
Anxiety improvement after 6 months | 6 months
  State-Trait Anxiety Index (STAI) Form-Y-1
Impulsiveness improvement after 6 months | 6 months
  Barratt Impulsiveness Scale
Self-rated Biochemical improvement after 6 months | 6 months
  Rosenberg Self-Biochemical Scale
Personality improvement after 6 months | 6 months
  Temperament and Character Inventory (TCI)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Amianto, MD, PhD, Principal Investigator — University of Torino; Secondo Fassino, MD, Study Chair — University of Torino
Locations (1):
- Villa Garda, Garda, Veneto, Italy

REFERENCES:
- [Derived] Brambilla F, Amianto F, Dalle Grave R, Fassino S. Lack of efficacy of psychological and pharmacological treatments of disorders of eating behavior: neurobiological background. BMC Psychiatry. 2014 Dec 24;14:376. doi: 10.1186/s12888-014-0376-7. PMID 25539757